CLINICAL TRIAL: NCT03761212
Title: Gait Parameters as Predictors of Functional and Activity Scores in Ankylosing Spondylitis : the FoLoMI Study
Brief Title: Function, Locomotion, Measurement and Inflammation
Acronym: FoLoMI
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC17.158.
Record Dates: First submitted 2018-07-19; First posted 2018-12-03 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing spondylitis; Gait; BASFI; BASDAI; 6MWT
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient with ankylosing spondylitis or axial spondyloarthritis: No intervention - observational study
- Healthy controls: Age and sex matched healthy controls

SUMMARY:
FoLoMI is a pilot study in which the investigators will seek to determine if gait spatio-temporal and kinematic parameters can explain the evolution of a functional score, the Bath Ankylosing Spondylitis Functional Index (BASFI), at 18 months.

The secondary objectives are: (1) to study the relationship between gait parameters measured at T0 and the BASFI at T0, (2) to study the relationship between gait parameters at T0 and the BASDAI at T0, (3) to assess general state of health of the patients and its evolution by appreciating: level of physical activity, state of fatigue, diurnal sleepiness and quality of life, and (4) to compare spatio-temporal gait parameters between patients and healthy controls.

DETAILED DESCRIPTION:
This longitudinal cohort study is aiming to follow 60 persons with ankylosing spondylitis during 18 months. Assessments will be conducted at baseline and every 6 months.

An healthy control group of 30 persons will be included and age and sex matched to the first 30 patients.

ELIGIBILITY:
Inclusion Criteria:

* Ankylosing spondylitis or Axial Spondyloarthritis patient
* Patient able to walk at least 180 meters without technical help
* Stable treatment for 3 months
* Affiliated to a social security system

Exclusion Criteria:

* Concomitant musculo-skeletal disease
* Cardio-respiratory disease with an impact on locomotion
* Hips, ankle or knee arthroplasty (scheduled or done within 18 months)
* No french understanding
* Central or peripheric neurologic disease
* Other disease with impact on posture, locomotion or prehension
* Quickly evolutive disease (less than 12 month life expectancy)
* Chemotherapy or radiotherapy ongoing
* Patient who live more than 50 km away from Grenoble Hospital
* Willing of pregnancy within 18 months
* People protected by law (Article L1121.5 of Public Health Code)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with Ankylosing Spondylitis or Axial Spondyloarthritis at any stage of disease evolution followed at the Rhumatology unit of Grenoble Hospital
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Gait speed | Baseline : Day 0
  Mean gait speed (m/s) will be assessed during a 10-m walk test at comfortable speed, under single and dual task, and its coefficient of variation calculate.
Stride time | Baseline : Day 0
  Mean stride time (s) will be assessed during a 10-m walk test at comfortable speed, under single and dual task, and its coefficient of variation calculate.
Stride length | Baseline : Day 0
  Mean stride length (m) will be assessed during a 10-m walk test at comfortable speed, under single and dual task, and its coefficient of variation calculate.
Double support time | Baseline : Day 0
  Double support time (%) will be assessed during a 10-m walk test at comfortable speed, under single and dual task, and its coefficient of variation calculate.
Stance time | Baseline : Day 0
  Stance time (%) will be assessed during a 10-m walk test at comfortable speed, under single and dual task, and its coefficient of variation calculate.
The Bath Ankylosing Spondylitis Functional Index (BASFI) | 18 months
  The self-administered Bath Ankylosing Functional Index (BASFI) measures functional consequences of ankylosing spondylitis (AS). The patient indicates its level of ability in ten domains of daily life: put the socks, bend to pick a pen from the floor, reach up to a high shelf, get up from a chair and from the floor, stand unsupported for 10 minutes, climb steps, look over the shoulder, do physically demanding activities and do a full days activities. Each question is answered on a 10 cm horizontal visual analog scale, the mean of which gives the BASFI score (0-10). Higher is the score, higher are the functional consequences of AS.

SECONDARY OUTCOMES:
Evolution of the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | From day 0 to 18-months
  The self-administered Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) measures disease activity. Six 10 cm horizontal visual analog scales are used to measure severity of fatigue, spinal and peripheral joint pain, localized tenderness and morning stiffness (qualitative and quantitative). The final BASDAI score has a range from 0 to 10, with higher scores meaning higher activity of the disease.
Evolution of the Bath Ankylosing Spondylitis Functional Index (BASFI) | From day 0 to 18-months
  The self-administered Bath Ankylosing Functional Index (BASFI) measures functional consequences of ankylosing spondylitis (AS). The patient indicates its level of ability in ten domains of daily life: put the socks, bend to pick a pen from the floor, reach up to a high shelf, get up from a chair and from the floor, stand unsupported for 10 minutes, climb steps, look over the shoulder, do physically demanding activities and do a full days activities. Each question is answered on a 10 cm horizontal visual analog scale, the mean of which gives the BASFI score (0-10). Higher is the score, higher are the functional consequences of AS.
Evolution of gait pattern | From day 0 to 18-months
  Gait pattern will be captured by Physilog sensors (Gait Up ®) and Opal sensors (APDM®) during a 10-m walk test in single and dual task, the iTUG and the i6MWT.
Evolution of physical activity | From day 0 to 18-months
  Patients will fill in the self-assessment questionnaire: International Physical Activity Questionnaires (IPAQ) to measure health-related physical activity. Data will be summarized according to each physical activity domain (walking, moderate and vigorous activities) and estimated time spend sitting per week. Then data will be used to estimate Metabolic Equivalent of Task (MET) energy expenditure assigned to each category.
Evolution of quality of life | From day 0 to 18-months
  Patients will fill in the self-assessment questionnaire: Short Form-36 (SF-36) to measure quality of life. Eight domains will be assessed : physical activity, daily life limitations, physical pain, health, social life, psychological health, psychological limitations, health evolution.
Evolution of daytime sleepiness | From day 0 to 18-months
  Patients will fill in the self-assessment questionnaire: Epworth score for evaluation of daytime sleepiness. Patients wil rate the chances that they would doze off or fall asleep while in eight different situations, from no chance to doze or sleep (0) to strong chance to sleep (3).
Evolution of tiredness | From day 0 to 18-months
  Patients will fill in the self-assessment questionnaire: Pichot score for evaluation of daytime tiredness. This scale assess the importance of tiredness to carry out daily activities.Patients rate how the eight proposals correspond to their feeling, from not at all (0) to extremely (4).
Evolution of lower limbs range of motion assessments | From day 0 to 18-months
  Lower limb range of motion will be assessed using a goniometer in each joint.
Evolution of foot function | From day 0 to 18-months
  Foot function will be assessed with the validated and commonly used Foot Function Index. Participants will rate 0 to 10 on a numeric scale, in 3 domains concerning feet, i.e. pain, disability and activity restriction. The score is out of 230 and translated out of 100. Higher scores are related to worse outcome.
Evolution of six minute walk distance | From day 0 to 18-months
  The instrumented six minute walk test (i6MWT) will be performed in a 30-m corridor.
Evolution of time to realize instrumented Timed Up and Go (iTUG) | From day 0 to 18-month
  Patients will performed the iTUG : they have to stand up from a chair, walk 7 meters, turn and go back to the chair, as fast as possible
Evolution of work impairment | From day 0 to 18-month
  The validated Work Productivity and Activity Impairment scale (WPAI) will be assessed to evaluate absenteeism, presenteeism, overall work productivity loss and activity impairment. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes.
Evolution of smoking status | From day 0 to 18-month
  Smoking status will be assessed with the calculation of number of pack-year smoked. It is calculated by multiplying the number of packs of cigarettes smoked per day by the number of years the person has smoked.
Evolution of nicotine dependence | From day 0 to 18-month
  Smoking status will be assessed with the validated and commonly used Fagerström index, giving a score from 0 to 10, with high scores related to high dependence
Evolution of social support | From day 0 to 18-month
  Social support will be assessed with the validated and commonly used Medical Outcome Study (MOS) Social Support Survey in French. The survey consists of four separate social support subscales and an overall functional social support index. A higher score for an individual scale or for the overall support index indicates more support.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Grenoble Alpes - hôpital sud, Échirolles, France

REFERENCES:
- [Background] Zochling J. Measures of symptoms and disease status in ankylosing spondylitis: Ankylosing Spondylitis Disease Activity Score (ASDAS), Ankylosing Spondylitis Quality of Life Scale (ASQoL), Bath Ankylosing Spondylitis Disease Activity Index (BASDAI), Bath Ankylosing Spondylitis Functional Index (BASFI), Bath Ankylosing Spondylitis Global Score (BAS-G), Bath Ankylosing Spondylitis Metrology Index (BASMI), Dougados Functional Index (DFI), and Health Assessment Questionnaire for the Spondylarthropathies (HAQ-S). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S47-58. doi: 10.1002/acr.20575. No abstract available. PMID 22588768
- [Background] Auvinet B, Chaleil D, Cabane J, Dumolard A, Hatron P, Juvin R, Lanteri-Minet M, Mainguy Y, Negre-Pages L, Pillard F, Riviere D, Maugars YM. The interest of gait markers in the identification of subgroups among fibromyalgia patients. BMC Musculoskelet Disord. 2011 Nov 11;12:258. doi: 10.1186/1471-2474-12-258. PMID 22078002
- [Background] Viccaro LJ, Perera S, Studenski SA. Is timed up and go better than gait speed in predicting health, function, and falls in older adults? J Am Geriatr Soc. 2011 May;59(5):887-92. doi: 10.1111/j.1532-5415.2011.03336.x. Epub 2011 Mar 15. PMID 21410448
- [Background] Del Din S, Carraro E, Sawacha Z, Guiotto A, Bonaldo L, Masiero S, Cobelli C. Impaired gait in ankylosing spondylitis. Med Biol Eng Comput. 2011 Jul;49(7):801-9. doi: 10.1007/s11517-010-0731-x. Epub 2011 Jan 13. PMID 21229328
- [Background] Verweij NM, Schiphorst AH, Pronk A, van den Bos F, Hamaker ME. Physical performance measures for predicting outcome in cancer patients: a systematic review. Acta Oncol. 2016 Dec;55(12):1386-1391. doi: 10.1080/0284186X.2016.1219047. Epub 2016 Oct 8. PMID 27718777
- [Background] Zebouni L, Helliwell PS, Howe A, Wright V. Gait analysis in ankylosing spondylitis. Ann Rheum Dis. 1992 Jul;51(7):898-9. doi: 10.1136/ard.51.7.898. PMID 1632666
- [Background] Mangone M, Scettri P, Paoloni M, Procaccianti R, Spadaro A, Santilli V. Pelvis-shoulder coordination during level walking in patients with ankylosing spondylitis. Gait Posture. 2011 May;34(1):1-5. doi: 10.1016/j.gaitpost.2011.02.002. Epub 2011 Mar 4. PMID 21377366
- [Result] Soulard J, Vaillant J, Baillet A, Gaudin P, Vuillerme N. The effects of a secondary task on gait in axial spondyloarthritis. Sci Rep. 2021 Oct 1;11(1):19537. doi: 10.1038/s41598-021-98732-z. PMID 34599222
- [Result] Soulard J, Vaillant J, Baillet A, Gaudin P, Vuillerme N. Gait and Axial Spondyloarthritis: Comparative Gait Analysis Study Using Foot-Worn Inertial Sensors. JMIR Mhealth Uhealth. 2021 Nov 9;9(11):e27087. doi: 10.2196/27087. PMID 34751663
- [Result] Soulard J, Vaillant J, Balaguier R, Vuillerme N. Spatio-temporal gait parameters obtained from foot-worn inertial sensors are reliable in healthy adults in single- and dual-task conditions. Sci Rep. 2021 May 13;11(1):10229. doi: 10.1038/s41598-021-88794-4. PMID 33986307
- [Result] Soulard J, Vaillant J, Balaguier R, Baillet A, Gaudin P, Vuillerme N. Foot-Worn Inertial Sensors Are Reliable to Assess Spatiotemporal Gait Parameters in Axial Spondyloarthritis under Single and Dual Task Walking in Axial Spondyloarthritis. Sensors (Basel). 2020 Nov 12;20(22):6453. doi: 10.3390/s20226453. PMID 33198119
- [Result] Soulard J, Vuillerme N, Gaudin P, Grange L, Baillet A, Cracowski JL, Juvin R, Vaillant J. Gait as predictor of physical function in axial spondyloarthritis: the prospective longitudinal FOLOMI (Function, Locomotion, Measurement, Inflammation) study protocol. Rheumatol Int. 2019 Oct;39(10):1681-1688. doi: 10.1007/s00296-019-04396-4. Epub 2019 Aug 7. PMID 31392500